CLINICAL TRIAL: NCT01750918
Title: An Open-Label, Four-Part, Phase I/II Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of the MEK Inhibitor GSK1120212, BRAF Inhibitor GSK2118436 and the Anti-EGFR Antibody Panitumumab in Combination in Subjects With BRAF-mutation V600E Positive Colorectal Cancer and in Subjects With CRC With Secondary Resistance to Prior Anti-EGFR Therapy
Brief Title: BRAF/MEK/EGFR Inhibitor Combination Study in Colorectal Cancer (CRC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116833; CDRB436C2201 (Other: Novartis); 2012-004802-81 (EudraCT Number)
Record Dates: First submitted 2012-12-06; First posted 2012-12-17 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-09

CONDITIONS: Cancer
Keywords: MEK inhibitor; anti-EGFR antibody; colorectal cancer; BRAF inhibitor
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms | interventions — dabrafenib; trametinib; Panitumumab

STUDY DESIGN:
Intervention Model Description: The original intention of the study was to include a randomized phase 2 portion of the study as a "Part 3"; however, a preliminary analysis did not meet predetermined criteria for efficacy. As a result, Part 3 of the study was not initiated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: Dabrafenib and Panitumumab (Experimental): In Part 1 subjects will be assigned to escalation cohort of the doublet of dabrafenib and panitumumab based on the monotherapy doses of dabrafenib (150 milligrams [mg] twice daily) and panitumumab (6 milligrams per kilogram [mg/kg] every-2-week [Q2W]). Dose escalation will follow a 3+3 dose escalation procedure. If the initial combination dose of dabrafenib and panitumumab in Cohort 1 (starting dose) is not tolerable, lower dose combination(s) may be evaluated.
  Interventions: Drug: Dabrafenib; Drug: Panitumumab
- Part 1: Dabrafenib, Trametinib and Panitumumab (Experimental): In Part 1 after the dabrafenib/panitumumab combination dose is defined, subsequent cohorts will evaluate the addition of trametinib based on a panitumumab dose that is one dose level lower than the dabrafenib/panitumumab dose defined in Cohort 1. Trametinib starting at 1.5 mg once daily will be added to the combination of dabrafenib and panitumumab. Dose escalation will follow a 3+3 dose escalation procedure until the full monotherapy doses of all agents are evaluated or the maximum tolerated dose is determined.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Panitumumab
- Part 2: Dabrafenib and panitumumab (Experimental): In Part 2, subjects will be assigned to expansion cohorts at a selected dose of dabrafenib in combination with panitumumab
  Interventions: Drug: Dabrafenib; Drug: Panitumumab
- Part 2: Dabrafenib, Trametinib and Panitumumab (Experimental): In Part 2, subjects will be assigned to expansion cohorts at selected dose of trametinib plus dabrafenib in combination with panitumumab.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Panitumumab
- Part 4a: Trametinib and Panitumumab (Experimental): Subject will be administered starting dose of Trametinib 2 mg once daily and Panitumumab 6mg/kg Q2W. If the initial combination dose of trametinib and panitumumab in Cohort 1 (starting dose) is not tolerable, the lower dose combination defined in de-escalation cohorts (Cohort -1A, -1B and/or -1C) may be evaluated. Cohort -1A: Trametinib 1.5 mg once daily and Panitumumab 6 mg/kg Q2W; Cohort -1B: Trametinib 2 mg once daily and Panitumumab 4.8 mg/kg Q2W; Cohort-1C: Trametinib 1.5 mg once daily and Panitumumab 4.8 mg/kg Q2W
  Interventions: Drug: Trametinib; Drug: Panitumumab
- Part 4b: Trametinib and Panitumumab (Experimental): In Part 4B cohort expansion, subjects will be assigned to expansion cohorts at a selected dose of trametinib in combination with panitumumab. Enrollment in expansion cohorts will be initiated once dose escalation for the trametinib /panitumumab combination has been completed. Subjects with advanced/metastatic CRC with either a BRAF-mutation (Cohort 1E) or who developed secondary resistance to prior anti-EGFR therapy (Cohort 2E).
  Interventions: Drug: Trametinib; Drug: Panitumumab
- Part 3a: Dabrafenib and Panitumumab (Experimental): Subjects will be randomized to receive dabrafenib plus panitumumab. Dose levels for dabrafenib, and panitumumab in Part 3 will be chosen based on emerging PK, PD, and tolerability data from Part 1 and Part 2.
  Interventions: Drug: Dabrafenib; Drug: Panitumumab
- Part 3b: Dabrafenib, Trametinib and Panitumumab (Experimental): Subjects will be randomized to receive study treatment as dabrafenib plus trametinib plus panitumumab. Dose levels for dabrafenib, trametinib and panitumumab in Part 3 will be chosen based on emerging PK, PD, and tolerability data from Part 1 and Part 2.
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Part 3c: Chemotherapy comparator (Experimental): Subjects will be randomized to receive chemotherapy comparator. The chemotherapy comparator will consist of a standard chemotherapy regimen with or without the addition of a biological agent, based on local practice preferences. The available chemotherapy regimens includes 5-fluorouracil-based chemotherapy
  Interventions: Device: 5-fluorouracil

INTERVENTIONS:
Drug: Dabrafenib — Each capsule contains 50 mg or 75 mg of GSK2118436; 50 mg strength capsules are Swedish orange (dark red) opaque hypromellose size 2 capsules and 75 mg strength capsules are pink opaque hypromellose size 1 capsules. The initial dosing regimen will be twice daily (BID) continuous oral daily dosing.
  Other Names: GSK2118436, DRB436
  Arms: Part 1: Dabrafenib and Panitumumab; Part 1: Dabrafenib, Trametinib and Panitumumab; Part 2: Dabrafenib and panitumumab; Part 2: Dabrafenib, Trametinib and Panitumumab; Part 3a: Dabrafenib and Panitumumab; Part 3b: Dabrafenib, Trametinib and Panitumumab
Drug: Trametinib — Each tablet contains 0.5mg or 2.0 mg GSK1120212; 0.5 mg is yellow modified oval biconvex film-coated tablets of size 4.8 mm X 8.9 mm and 2 mg as pink round biconvex film coated tablets;7.5 mm in diameter. The initial dosing regimen will be once daily continuous oral daily dosing.
  Other Names: GSK1120212, TMT212
  Arms: Part 1: Dabrafenib, Trametinib and Panitumumab; Part 2: Dabrafenib, Trametinib and Panitumumab; Part 3b: Dabrafenib, Trametinib and Panitumumab; Part 4a: Trametinib and Panitumumab; Part 4b: Trametinib and Panitumumab
Drug: Panitumumab — Panitumumab is a sterile, colorless, translucent-to-white amorphous, proteinaceous powder available as 100 mg panitumumab in 5 mL (20 mg/mL) single-use vial; 200 mg panitumumab in 10 mL (20 mg/mL) single-use vial; 400 mg panitumumab in 20 mL (20 mg/mL) single-use vial; to be administered as an intravenous infusion over 60 minutes, every 14 days. Doses higher than 1000 mg should be administered over 90 minutes.
  Arms: Part 1: Dabrafenib and Panitumumab; Part 1: Dabrafenib, Trametinib and Panitumumab; Part 2: Dabrafenib and panitumumab; Part 2: Dabrafenib, Trametinib and Panitumumab; Part 3a: Dabrafenib and Panitumumab; Part 4a: Trametinib and Panitumumab; Part 4b: Trametinib and Panitumumab
Device: 5-fluorouracil — 5-fluorouracil-based chemotherapy
  Arms: Part 3c: Chemotherapy comparator

SUMMARY:
This was a four part, phase I/II study aimed to evaluate the safety, tolerability and efficacy of combination of an anti-EGFR antibody panitumumab (P) either with a BRAF inhibitor (dabrafenib (D); GSK2118436) alone or with the combination of a BRAF inhibitor and a MEK inhibitor (trametinib (T); GSK1120212) in patients with BRAF-mutant V600E advanced or mCRC. The goal was to: 1) Determine RP2R/MTD for doublet (D+P) and triplet (D+T+P) combinations in Part 1; 2) Assess clinical activity for these combinations in Part 2; 3) Determine RP2R/MTD for double (T+P) combination in Part 4A, and assess clinical activity of this combination in two patient populations in Part 4B (patients with BRAF-V600E mutation-positive advanced or metastatic CRC and patients with advanced or metastatic CRC with secondary resistance to anti-EGFR therapy).

DETAILED DESCRIPTION:
Part 1: Dose escalation This was a dose escalation part intended to evaluate safety, tolerability, PK, PD, clinical activity and determine RP2R/MTD for the doublet (D+P) and the triplet (D+T+P) combinations in patients with BRAF-mutation V600E positive advanced or metastatic CRC. A 3+3 dose escalation procedure was followed. Dosing for dabrafenib and trametinib was continuous daily dosing while panitumumab was dosed once every two weeks (Q2W). Patients were evaluated for dose-limiting toxicities (DLTs) during the first 28 days of treatment.

Part 2A:

This was a cohort expansion part to assess the safety and preliminary clinical activity of the optimal safe and tolerable dose combinations (D+P)/(D+T+P) defined in Part 1.

Part 2B:

In this part, additional patients were enrolled into the triplet (D+T+P) combination at two dose levels in to further explore safety, tolerability and clinical activity. Up to 10 patients each with no prior treatment (First Line Population), and up to 20 patients each with at least one prior treatment (Second to Fourth Line Population) were planned to be enrolled in dose Cohorts 3A and 4.

Part 3: Randomized Phase 2 Study The randomized phase 2 portion (Phase 3) of the study was not pursued as the observed responses in any of the cohorts did not meet the predefined criteria at the time of the preliminary analysis (data cut-off date: 06-May-2016).

Part 4 This part was designed to identify the RP2R/MTD and initial clinical activity for the doublet (T+P) combination in patients BRAF-mutation V600E positive advanced or metastatic CRC, and advanced or metastatic CRC with secondary resistance to prior anti-EGFR therapy.

Part 4A: Dose Escalation This was a dose escalation part intended to determine RP2R/MTD for the doublet (T+P) combination in patients with BRAF-mutation V600E positive advanced or metastatic CRC. Approximately 18 patients (~6 each cohort) were planned to be enrolled in Part 4A. A 3+3 dose escalation procedure was followed. Dosing for trametinib was continuous daily dosing while panitumumab was dosed once every two weeks (Q2W). Patients were evaluated for DLTs during the first 28 days of treatment.

Part 4B: Cohort Expansion This was a cohort expansion part intended to evaluate safety and efficacy of the doublet (T+P) combination. Up to 20 patients in each of two expansion cohorts were planned to be enrolled at the starting dose cohort or MTD from Part 4A.

ELIGIBILITY:
Inclusion Criteria: Subjects eligible for enrolment in this study must meet all of the following criteria

* Provided written informed consent,
* Male or female >=18 years of age and able to swallow and retain orally administered study treatment and does not have any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
* Part 1 and Part 2: Histologically- or cytologically-confirmed diagnosis of advanced or metastatic BRAF V600E mutation positive CRC
* Part 4A and 4B ONLY: Histologically- or cytologically-confirmed diagnosis of advanced or metastatic CRC that either harbours the BRAF V600E -mutation, as determined by relevant genetic testing OR has developed secondary resistance to anti-EGFR therapy, defined as patients that derived benefit (disease control based on investigator assessment for >6 months OR partial response [confirmed or unconfirmed] based on RECIST 1.1) from prior anti-EGFR-containing therapy (as defined below) and then subsequently progressed on therapy. The anti-EGFR therapy must have been the most recent therapy and the patient must have progressed based on investigator assessment within 3 months of screening. Acceptable prior anti-EGFR-containing therapies include: a. Monotherapy anti-EGFR, including cetuximab or panitumumab OR b. irinotecan/anti-EGFR combo after previously having disease progression (based on investigator assessment) on an irinotecan-containing regimen
* Part 3: Histologically- or cytologically-confirmed diagnosis of BRAFV600E mutation positive advanced or metastatic colorectal cancer (CRC who are eligible to receive fluoropyrimidine-containing chemotherapy regimen that have experienced documented radiographic progression on one prior line of fluoropyrimidine-containing chemotherapy (previous anti-EGFR therapy is excluded), Second-line for advanced/metastatic disease, having failed or been intolerant to at least one regimen of fluoropyrimidine-containing chemotherapy including irinotecan or oxaliplatin in the advanced/metastatic setting. Enrollment in Part 3 may only occur following confirmation of KRAS wild-type cancer.
* Archival tissue is required; if archival tissue is not available or found to not contain tumor tissue, a fresh biopsy is required.
* Measurable disease per RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use one of the contraception methods listed in protocol.
* Female subjects are eligible if: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal female defined as 12 months of spontaneous amenorrhea to be verified with a follicle-stimulating hormone (FSH) level >40 Milli-international units per milliliter (MIU/mL) and estradiol level <40 picogram per milliliter (pg/mL). Child-bearing potential and agrees to use one of the contraceptive methods listed in protocol.
* Female subjects must agree to use contraception from 7 days prior to the first dose of study drug(s) until 6 months after the last dose of panitumumab, until 4 months after the last dose of trametinib, or 4 weeks after the last dose of dabrafenib, whichever is longer. Additionally, women of childbearing potential must have had a negative serum pregnancy test within 7 days prior to the first dose of study drug(s).
* Adequate organ system function as defined in absolute neutrophil count greater than or equal to 1.2X10^9/Liter (L), hemoglobin greater than or equal to 9 grams per deciliter (g/dL) or 5.6 millimoles per litre (mmol/L), platelets greater than or equal to 75 × 10^9/L, Prothrombin Time / International Normalized Ratio (PT/INR) and Partial Thromboplastin Time (PTT) less than or equal to 1.5X upper limit of normal (ULN); serum magnesium greater than or equal to the lower limit of normal (LLN); albumin greater than or equal to 2.5 g/dL or 25 grams per liter (g/L), total bilirubin less than or equal to 1.5XULN, and Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) less than or equal to 2.5X ULN; creatinine less than or equal to 1.5XULN or calculated creatinine clearance greater than or equal to 50mL/min; left ventricular ejection fraction (LVEF) greater than or equal to the LLN by echocardiography (ECHO) or multigated acquisition scan (MUGA).
* Subjects enrolled in France or Italy: In France or Italy, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria: Subjects meeting any of the following criteria must not be enrolled in the study

* History of prior malignancy, other than colorectal cancer.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator's assessment).
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy or biologic therapy).
* Prior exposure to a MEK inhibitor.
* Part 1, Part 2 and BRAF-mutant patients in Part 4 ONLY: Prior exposure to a BRAF inhibitor.
* Part 1, Part 2 and BRAF-mutant patients in Part 4 ONLY: Known presence of KRAS-mutation based on previous KRAS-testing. Note: Prospective KRAS testing is not required. However, if the results of previous KRAS testing are known, they must be used in assessing eligibility. KRAS testing will be performed retrospectively for all patients.
* Part 3: Prior exposure to EGFR inhibitors or an anti-EGFR antibody
* Received an investigational or approved anti-cancer drug within 4 weeks, or within 5 half-lives (whichever is shorter) of the first dose of study drug(s). At least 14 days must have passed between the last dose of prior investigational agent and the first dose of study drug(s).
* Part 3: Received more than one prior anti-cancer therapy in the metastatic setting, exclusive of previous adjuvant regimens. Previous investigational anti-cancer therapy in the metastatic setting is prohibited.
* Current use of a prohibited medication or requirement to dose with any of these medications during treatment with study drug(s).
* Known Hepatitis B, or Hepatitis C infection.
* Any major surgery, radiotherapy or immunotherapy within the 4 weeks prior to first dose of study drug(s). Limited radiotherapy with in the 2 weeks prior to first dose of study drug(s).
* Chemotherapy regimens with delayed toxicity within the 3 weeks prior to first dose of study drug(s). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within 2 weeks prior to first dose of study drug(s).
* Unresolved toxicity greater than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4 Grade 1 from previous anti-cancer therapy, with the exception of Grade 2 alopecia, Grade 2 neuropathy, or laboratory values that are allowed per inclusion criteria.
* History of retinal vein occlusion (RVO).
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism or excretion of drugs. Previous colectomy is acceptable.
* Subjects with brain metastases are excluded, unless: All known lesions must be previously treated with surgery or stereotactic radio-surgery, and Brain lesion(s), if present, must be confirmed stable (i.e., no increase in lesion size) for >=90 days prior to first dose of study drug(s). This must be documented with two consecutive MRI or CT scans using contrast, and Asymptomatic with no corticosteroids requirement for >=30 days prior to first dose of study drug(s), and No enzyme-inducing anticonvulsants for >=14 days prior to first dose of study drug(s). In addition, for subjects that had brain metastases but currently have no evidence of disease (NED), NED for >=12 weeks is required and must be confirmed by two consecutive MRI or CT scans (using contrast) separated by >=6 weeks, prior to randomization. Enrollment of a subject with brain metastases who meet the above criteria requires approval of a GlaxoSmithKline (GSK) Medical Monitor.
* Psychological, familial, sociological or geographical conditions that do not permit compliance with the protocol.
* History or evidence of cardiovascular risk including any of the following: LVEF<LLN; A QT interval corrected for heart rate using the Bazett's formula (QTcB;) ≥ 480 milliseconds (msec);.History or evidence of current clinically significant uncontrolled arrhythmias. Exception: Subjects with controlled atrial fibrillation for >30 days prior to randomization are eligible. History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization. History or evidence of current >= Class II congestive heart failure as defined by New York Heart Association (NYHA). Treatment refractory hypertension defined as a blood pressure of systolic> 140 millimeter of mercury (mm Hg) and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy; Subjects with intra-cardiac defibrillators or permanent pacemakers; Known cardiac metastases
* Unstable pulmonary embolism, deep vein thrombosis, or other significant arterial/venous thromboembolic event <=30 days before randomization. If on anticoagulation, subject must be on stable therapeutic dose prior to randomization.
* Subjects with a history of pneumonitis or interstitial lung disease (ILD).
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drug(s) or their excipients.
* Pregnant or lactating female.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Uncontrolled diabetes or other medical condition that may interfere with assessment of toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (7):
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Italy (2):
  - Novartis Investigative Site, Candiolo
  - Novartis Investigative Site, Milan
- Japan (2):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Chiba
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Barcelona, Spain
- Novartis Investigative Site, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
This product has been acquired by Novartis Pharmaceuticals. Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 20 study centers across eight countries: Belgium (2), France (2), Italy (2), Japan (2), Netherlands (2), Spain (1), UK (1) and USA (8).
Pre-assignment Details: Since the tumor type enrolled in Part 1 and Part 2 was the same (metastatic colorectal cancer), the results were summarized by combination groups (and not by study parts) to allow a more meaningful interpretation of study results based on dose
Groups:
- Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W: Part 1+2A+2B - Triple combination (Trametinib + Dabrafenib + Panitumumab): Dabrafenib 150 mg BID + Trametinib 1.5 mg QD + Panitumumab 4.8 mg/kg Q2W
- Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W: Part 1+2A+2B - Triple combination (Trametinib + Dabrafenib + Panitumumab): Dabrafenib 150 mg BID + Trametinib 1.5 mg QD + Panitumumab 6.0 mg/kg Q2W
- Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W: Part 1+2A+2B - Triple combination (Trametinib + Dabrafenib + Panitumumab): Dabrafenib 150 mg BID + Trametinib 2.0 mg QD + Panitumumab 4.8 mg/kg Q2W
- Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W: Part 1+2A+2B - Triple combination (Trametinib + Dabrafenib + Panitumumab): Dabrafenib 150 mg BID + Trametinib 2.0 mg QD + Panitumumab 6.0 mg/kg Q2W
- Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab): Trametinib 2.0 mg QD + Panitumumab 6.0 mg/kg Q2W
- Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab): Trametinib 1.5 mg QD + Panitumumab 6.0 mg/kg Q2W
- Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab): Trametinib 2.0 mg QD + Panitumumab 4.8 mg/kg Q2W
- Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W: Part 1+2A - Double combination (Dabrafenib + Panitumumab): Dabrafenib 150 mg BID + Panitumumab 6.0 mg/kg Q2W
Period: Overall Study
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Started (All patients who were treated with at least one dose of the study drug at the time of the final analysis.) | 3 | 4 | 36 | 50 | 13 | 20 | 20 | 20
Pharmacokinetic Population (All patients in the All Treated Population for whom a PK sample was obtained and analyzed.) | 3 | 4 | 35 | 48 | 12 | 19 | 18 | 20
Biomarker Population (All patients in the All Treated Population whom a tumor biopsy/tissue was obtained and analyzed.) | 3 | 4 | 36 | 50 | 13 | 17 | 19 | 20
Crossover Population (Subset of patients in double combination who crossed over to triplet combination.) | 0 | 0 | 0 | 0 | 4 | 2 | 5 | 5
Completed | 3 | 4 | 28 | 44 | 12 | 17 | 17 | 16
Not Completed | 0 | 0 | 8 | 6 | 1 | 3 | 3 | 4
Not completed — Last patient transitioned to a rollover protocol | 0 | 0 | 5 | 2 | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Since, BRAF V600 mutant patients (MBRAF population) and KRAS wildtype patients progressing after EGFR based therapy (anti-EGFR population) were categorized as biologically distinct populations, doublet combination Trametinib + Panitumumab (T+P) was split into MBRAF and anti-EGFR patients for Baseline Characteristics and efficacy analysis to allow a more meaningful interpretation of study results.
Groups:
- Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab) mBRAF Patients: Trametinib 2.0 mg QD + Panitumumab 6.0 mg/kg Q2W
- Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab) mBRAF Patients: Trametinib 1.5 mg QD + Panitumumab 6.0 mg/kg Q2W
- Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab) mBRAF Patients: Trametinib 2.0 mg QD + Panitumumab 4.8 mg/kg Q2W
- Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab) anti-EGFR Patients: Trametinib 2.0 mg QD + Panitumumab 6.0 mg/kg Q2W
- Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab) anti-EGFR Patients: Trametinib 1.5 mg QD + Panitumumab 6.0 mg/kg Q2W
- Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W: Part 4A+4B - Double combination (Trametinib + Panitumumab) anti-EGFR: Trametinib 2.0 mg QD + Panitumumab 4.8 mg/kg Q2W
- Total: Total of all reporting groups
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W | Total
Number analyzed (Participants) | 3 | 4 | 36 | 50 | 11 | 10 | 10 | 2 | 10 | 10 | 20 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 20 | 30 | 8 | 6 | 9 | 2 | 9 | 6 | 12 | 108
  >=65 years | 1 | 0 | 16 | 20 | 3 | 4 | 1 | 0 | 1 | 4 | 8 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 21 | 33 | 5 | 7 | 6 | 0 | 3 | 3 | 11 | 94
  Male | 0 | 2 | 15 | 17 | 6 | 3 | 4 | 2 | 7 | 7 | 9 | 72
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 3 | 4 | 28 | 37 | 10 | 7 | 7 | 2 | 8 | 10 | 18 | 134
  Black or African American | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
  Asian | 0 | 0 | 7 | 9 | 1 | 2 | 3 | 0 | 2 | 0 | 1 | 25
  Missing | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group Performance Status (ECOG PS) score classifies participants according to their functional impairment, with scores ranging from 0 (fully active) to 5 (dead). ECOG PS: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    Grade 0 | 2 | 2 | 17 | 27 | 6 | 5 | 6 | 2 | 5 | 8 | 13 | 93
    Grade 1 | 1 | 2 | 19 | 23 | 5 | 5 | 4 | 0 | 5 | 2 | 7 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The distribution of adverse events was done via the analysis of frequencies for Adverse Events, Serious Adverse Events and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters. Only descriptive analysis performed.
Time Frame: From study treatment start date till 30 days safety follow-up, assessed up to approximately 90 months
Population: All treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 36 | 50 | 13 | 20 | 20 | 20
Participants
  Any Adverse Event (AE) | 3 | 4 | 36 | 50 | 13 | 20 | 20 | 20
  AEs related to study treatment | 3 | 4 | 36 | 49 | 13 | 19 | 20 | 20
  AEs leading to permanent discontinuation of study treatment | 0 | 0 | 9 | 12 | 3 | 4 | 2 | 1
  AEs leading to dose reduction | 2 | 2 | 19 | 37 | 7 | 14 | 14 | 5
  AEs leading to dose interruption/delay | 2 | 4 | 32 | 43 | 9 | 15 | 18 | 9
  Any serious adverse event (SAE) | 2 | 2 | 21 | 28 | 6 | 10 | 9 | 6
  SAEs related to study treatment | 1 | 1 | 12 | 18 | 5 | 4 | 5 | 5
  Fatal SAEs | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Fatal SAEs related to study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Deaths during treatment period | 0 | 0 | 3 | 2 | 1 | 2 | 0 | 0
  Deaths during follow-up period | 3 | 4 | 25 | 42 | 11 | 15 | 17 | 16

2. Primary Outcome: Overall Response Rate (ORR)
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) was used for efficacy based on radiological assessment of tumor burden: CR = Complete Response, disappearance of all target lesions; PR = Partial Response, >=30% decrease in the sum of the longest diameter of target lesions; PD = progressive disease, >=20% increase in sum of target lesions and/or presence of new lesions and/or substantial increase in non-target lesion; SD = stable disease, response not meeting CR or PR or PD; ORR = overall response rate, defined as CR+PR
Time Frame: From study treatment start date until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 90 months
Population: All treated population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 36 | 50 | 11 | 10 | 10 | 2 | 10 | 10 | 20
Percentage of Participants | 67 [9.4 to 99.2] | 0 [0.0 to 60.2] | 28 [14.2 to 45.2] | 20 [10.0 to 33.7] | 0 [0.0 to 28.5] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 0 [0.0 to 84.2] | 0 [0.0 to 30.8] | 0 [0.0 to 30.8] | 10 [1.2 to 31.7]

3. Primary Outcome: Part 3: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) was defined as the time from study treatment start date to the date of first radiologically documented progression or death due to any cause. If a patient did not progress or die at the time of the analysis data cut-off or start of new antineoplastic therapy, PFS was censored at the date of the last adequate tumor assessment before the earliest of the cut-off date or the start date of additional anti-neoplastic therapy. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria RECIST v1.1, as 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline and/or unequivocal progression of the non-target lesions and/or appearance of a new lesion. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 2
Population: All treated population. The original intention of the study was to include a randomized phase 2 portion of the study as a "Part 3"; however, a preliminary analysis did not meet predetermined criteria for efficacy. As a result, Part 3 of the study was not initiated.
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) was defined as the time from the first documented occurrence of response (PR or CR) until the date of the first documented progression based on RECIST v1.1 or death.
Time Frame: as for outcome 2
Population: All treated population. Only participants with an evaluable DoR events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 1 | 0 | 7 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Months | 2.9 [NA to NA] — Only 1 participant analyzed |  | 8.9 [2.8 to NA] — Upper limit 95% CI interval not estimable due to insufficient number of participants with events. | 6.9 [2.7 to 63.1] |  |  |  |  |  |  | 6.9 [5.9 to 8.0]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 3
Time Frame: as for outcome 2
Population: All treated population. Only participants with an evaluable PFS events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 2 | 4 | 25 | 41 | 10 | 10 | 10 | 2 | 9 | 9 | 19
Months | 8.3 [4.1 to 12.6] | 4.0 [2.1 to 11.0] | 7.4 [3.1 to 10.0] | 4.2 [3.0 to 5.2] | 2.9 [1.3 to 4.2] | 1.6 [0.4 to 2.9] | 2.7 [1.2 to 2.8] | 3.0 [2.8 to 3.2] | 2.8 [1.3 to 4.2] | 2.9 [1.3 to 3.6] | 3.5 [2.8 to 5.8]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time to death due to any cause.
Time Frame: From study treatment start date until date of of death from any cause, assessed up to approximately 90 months
Population: All treated population. Only participants with an evaluable OS events were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 28 | 44 | 10 | 9 | 9 | 2 | 8 | 8 | 16
Months | 20.7 [4.9 to 58.6] | 14.7 [4.1 to 46.4] | 18.8 [8.1 to 20.8] | 8.3 [7.2 to 10.2] | 8.2 [2.3 to 12.8] | 5.8 [2.3 to 7.2] | 8.6 [5.4 to 16.7] | 11.2 [10.6 to 11.8] | 11.5 [5.8 to 39.8] | 19.9 [2.9 to 35.9] | 13.9 [6.7 to 22.0]

7. Secondary Outcome: Cmax of Dabrafenib and Derived Metabolites in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Maximum observed concentration (Cmax) of Dabrafenib and derived metabolites were listed and summarized using descriptive statistics.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: Pharmacokinetic population. Only participants with an evaluable PK sample collected at each timepoint were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 8 | 22
ng/mL
  Dabrafenib @ D1 (n=3,4,8,22) | 2440 (91.3) | 2400 (162.8) | 2180 (83.6) | 1550 (87.2)
  Dabrafenib @ D15 (n=1,3,5,18): number analyzed (Participants) | 1 | 3 | 5 | 18
  Dabrafenib @ D15 (n=1,3,5,18) | 2410 (NA) — Only one participant analyzed | 1800 (161.7) | 1100 (331.5) | 1580 (84.3)
  Dabrafenib @ Wk8 (n=0,0,0,2): number analyzed (Participants) | 0 | 0 | 0 | 2
  Dabrafenib @ Wk8 (n=0,0,0,2) |  |  |  | 699 (237.8)
  Dabrafenib @ Wk12 (n=0,0,0,3): number analyzed (Participants) | 0 | 0 | 0 | 3
  Dabrafenib @ Wk12 (n=0,0,0,3) |  |  |  | 848 (3137.6)
  Dabrafenib @ Wk16 (n=0,1,0,1): number analyzed (Participants) | 0 | 1 | 0 | 1
  Dabrafenib @ Wk16 (n=0,1,0,1) |  | 74.1 (NA) — Only one participant analyzed |  | 2150 (NA) — Only one participant analyzed
  Dabrafenib @ Wk20 (n=0,1,1,1): number analyzed (Participants) | 0 | 1 | 1 | 1
  Dabrafenib @ Wk20 (n=0,1,1,1) |  | 136 (NA) — Only one participant analyzed | 7.92 (NA) — Only one participant analyzed | 5700 (NA) — Only one participant analyzed
  GSK2167542 @ D1 (n=3,4,7,21): number analyzed (Participants) | 3 | 4 | 7 | 21
  GSK2167542 @ D1 (n=3,4,7,21) | 120 (43.4) | 21.2 (109.0) | 34.8 (76.6) | 23.3 (97.8)
  GSK2167542 @ D15 (n=1,3,5,19): number analyzed (Participants) | 1 | 3 | 5 | 19
  GSK2167542 @ D15 (n=1,3,5,19) | 311 (NA) — Only one participant analyzed | 360 (77.0) | 347 (94.5) | 328 (70.9)
  GSK2167542 @ Wk8 (n=1,2,0,3): number analyzed (Participants) | 1 | 2 | 0 | 3
  GSK2167542 @ Wk8 (n=1,2,0,3) | 266 (NA) — Only one participant analyzed | 312 (88.8) |  | 197 (47.3)
  GSK2167542 @ Wk12 (n=1,2,0,3): number analyzed (Participants) | 1 | 2 | 0 | 3
  GSK2167542 @ Wk12 (n=1,2,0,3) | 132 (NA) — Only one participant analyzed | 130 (23.7) |  | 385 (86.0)
  GSK2167542 @ Wk16 (n=2,2,0,2): number analyzed (Participants) | 2 | 2 | 0 | 2
  GSK2167542 @ Wk16 (n=2,2,0,2) | 209 (65.2) | 135 (79.4) |  | 421 (106.9)
  GSK2167542 @ Wk20 (n=0,2,1,2): number analyzed (Participants) | 0 | 2 | 1 | 2
  GSK2167542 @ Wk20 (n=0,2,1,2) |  | 269 (110.5) | 82.1 (NA) — Only one participant analyzed | 404 (131.2)
  GSK2285403 @ D1 (n=3,4,8,22) | 1430 (51.4) | 1010 (92.4) | 1060 (56.6) | 674 (71.0)
  GSK2285403 @ D15 (n=1,3,5,19): number analyzed (Participants) | 1 | 3 | 5 | 19
  GSK2285403 @ D15 (n=1,3,5,19) | 1050 (NA) — Only one participant analyzed | 718 (69.6) | 477 (202.1) | 656 (86.0)
  GSK2285403 @ Wk8 (n=1,2,0,3): number analyzed (Participants) | 1 | 2 | 0 | 3
  GSK2285403 @ Wk8 (n=1,2,0,3) | 32.4 (NA) — Only one participant analyzed | 221 (6687.0) |  | 238 (310.1)
  GSK2285403 @ Wk12 (n=1,2,0,3): number analyzed (Participants) | 1 | 2 | 0 | 3
  GSK2285403 @ Wk12 (n=1,2,0,3) | 21.4 (NA) — Only one participant analyzed | 21.3 (2.7) |  | 518 (362.8)
  GSK2285403 @ Wk16 (n=2,2,0,2): number analyzed (Participants) | 2 | 2 | 0 | 2
  GSK2285403 @ Wk16 (n=2,2,0,2) | 59.4 (358.1) | 42.5 (59.0) |  | 200 (2064.4)
  GSK2285403 @ Wk20 (n=0,2,1,2): number analyzed (Participants) | 0 | 2 | 1 | 2
  GSK2285403 @ Wk20 (n=0,2,1,2) |  | 46.4 (189.2) | 12 (NA) — Only one participant analyzed | 284 (812.1)

8. Secondary Outcome: Cmax of Trametinib in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Maximum observed concentration (Cmax) of Trametinib was listed and summarized using descriptive statistics.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 8 | 22
ng/mL
  Day 1 (n=3,4,8,22) | 5.31 (28.6) | 5.08 (82.8) | 10.3 (58.5) | 4.65 (112.4)
  Day 15 (n=1,3,4,18): number analyzed (Participants) | 1 | 3 | 4 | 18
  Day 15 (n=1,3,4,18) | 24 (NA) — Only one participant analyzed | 20 (33.1) | 22.2 (42.9) | 19.5 (47.6)
  Week 8 (n=2,0,0,2): number analyzed (Participants) | 2 | 0 | 0 | 2
  Week 8 (n=2,0,0,2) | 9.2 (54.6) |  |  | 30.1 (18.2)
  Week 12 (n=2,0,0,3): number analyzed (Participants) | 2 | 0 | 0 | 3
  Week 12 (n=2,0,0,3) | 6.2 (67.1) |  |  | 19.7 (73.2)
  Week 16 (n=1,1,0,1): number analyzed (Participants) | 1 | 1 | 0 | 1
  Week 16 (n=1,1,0,1) | 12.4 (NA) — Only one participant analyzed | 11.2 (NA) — Only one participant analyzed |  | 29.5 (NA) — Only one participant analyzed
  Week 20 (n=1,0,1,1): number analyzed (Participants) | 1 | 0 | 1 | 1
  Week 20 (n=1,0,1,1) | 11.3 (NA) — Only one participant analyzed |  | 6.89 (NA) — Only one participant analyzed | 38.1 (NA) — Only one participant analyzed

9. Secondary Outcome: Tmax of Dabrafenib and Derived Metabolites in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Time of occurrence of Cmax (tmax) of Dabrafenib and derived metabolites were listed and summarized using descriptive statistics.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 8 | 22
Hour (hr)
  Dabrafenib @ D1 (n=3,4,8,22) | 2 [1 to 4] | 1.5 [1 to 4] | 2 [1 to 4] | 2 [1 to 8]
  Dabrafenib @ D15 (n=1,3,5,18): number analyzed (Participants) | 1 | 3 | 5 | 18
  Dabrafenib @ D15 (n=1,3,5,18) | 2.05 [2.05 to 2.05] | 2 [1 to 2] | 1 [0 to 1.55] | 2 [1 to 6]
  Dabrafenib @ Wk8 (n=0,0,0,2): number analyzed (Participants) | 0 | 0 | 0 | 2
  Dabrafenib @ Wk8 (n=0,0,0,2) |  |  |  | 4.75 [1.92 to 7.58]
  Dabrafenib @ Wk12 (n=0,0,0,3): number analyzed (Participants) | 0 | 0 | 0 | 3
  Dabrafenib @ Wk12 (n=0,0,0,3) |  |  |  | 4.88 [0.92 to 11]
  Dabrafenib @ Wk16 (n=0,1,0,1): number analyzed (Participants) | 0 | 1 | 0 | 1
  Dabrafenib @ Wk16 (n=0,1,0,1) |  | 11.5 [11.5 to 11.5] |  | 2.23 [2.23 to 2.23]
  Dabrafenib @ Wk20 (n=0,1,1,1): number analyzed (Participants) | 0 | 1 | 1 | 1
  Dabrafenib @ Wk20 (n=0,1,1,1) |  | 12 [12 to 12] | 0.42 [0.42 to 0.42] | 0.87 [0.87 to 0.87]
  GSK2167542 @ D1 (n=3,4,7,21): number analyzed (Participants) | 3 | 4 | 7 | 21
  GSK2167542 @ D1 (n=3,4,7,21) | 8 [4 to 8] | 7 [6 to 8] | 8 [4 to 8] | 8 [4 to 8]
  GSK2167542 @ D15 (n=1,3,5,19): number analyzed (Participants) | 1 | 3 | 5 | 19
  GSK2167542 @ D15 (n=1,3,5,19) | 6.03 [6.03 to 6.03] | 1 [0 to 2] | 2 [0.82 to 6] | 2 [0 to 32]
  GSK2167542 @ Wk8 (n=1,2,0,3): number analyzed (Participants) | 1 | 2 | 0 | 3
  GSK2167542 @ Wk8 (n=1,2,0,3) | 16.8 [16.8 to 16.8] | 16 [15.8 to 16.3] |  | 7.58 [1.92 to 13.3]
  GSK2167542 @ Wk12 (n=1,2,0,3): number analyzed (Participants) | 1 | 2 | 0 | 3
  GSK2167542 @ Wk12 (n=1,2,0,3) | 16.3 [16.3 to 16.3] | 16.6 [16.5 to 16.7] |  | 4.88 [0.92 to 11]
  GSK2167542 @ Wk16 (n=2,2,0,2): number analyzed (Participants) | 2 | 2 | 0 | 2
  GSK2167542 @ Wk16 (n=2,2,0,2) | 21.3 [14.7 to 27.8] | 14.4 [11.5 to 17.3] |  | 7.87 [2.23 to 13.5]
  GSK2167542 @ Wk20 (n=0,2,1,2): number analyzed (Participants) | 0 | 2 | 1 | 2
  GSK2167542 @ Wk20 (n=0,2,1,2) |  | 14.5 [12 to 17] | 0.42 [0.42 to 0.42] | 7.35 [0.87 to 13.8]
  GSK2285403 @ D1 (n=3,4,3,22): number analyzed (Participants) | 3 | 4 | 3 | 22
  GSK2285403 @ D1 (n=3,4,3,22) | 4 [2 to 6] | 3 [2 to 4] | 3 [2 to 6] | 4 [1 to 8]
  GSK2285403 @ D15 (n=1,3,5,19): number analyzed (Participants) | 1 | 3 | 5 | 19
  GSK2285403 @ D15 (n=1,3,5,19) | 4 [4 to 4] | 2 [1 to 4] | 1 [0 to 2.02] | 2.02 [1.67 to 32]
  GSK2285403 @ Wk8 (n=1,2,0,3): number analyzed (Participants) | 1 | 2 | 0 | 3
  GSK2285403 @ Wk8 (n=1,2,0,3) | 16.8 [16.8 to 16.8] | 16 [15.8 to 16.3] |  | 7.58 [1.92 to 13.3]
  GSK2285403 @ Wk12 (n=1,2,0,3): number analyzed (Participants) | 1 | 2 | 0 | 3
  GSK2285403 @ Wk12 (n=1,2,0,3) | 16.3 [16.3 to 16.3] | 16.6 [16.5 to 16.7] |  | 4.88 [0.92 to 11]
  GSK2285403 @ Wk16 (n=2,2,0,2): number analyzed (Participants) | 2 | 2 | 0 | 2
  GSK2285403 @ Wk16 (n=2,2,0,2) | 21.3 [14.7 to 27.8] | 14.4 [11.5 to 17.3] |  | 7.87 [2.23 to 13.5]
  GSK2285403 @ Wk20 (n=0,2,1,2): number analyzed (Participants) | 0 | 2 | 1 | 2
  GSK2285403 @ Wk20 (n=0,2,1,2) |  | 14.5 [12 to 17] | 0.42 [0.42 to 0.42] | 7.35 [0.87 to 13.8]

10. Secondary Outcome: Tmax of Trametinib in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Time of occurrence of Cmax (tmax) of Trametinib was listed and summarized using descriptive statistics.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 8 | 22
Hour (hr)
  Day 1 (n=3,4,8,22) | 1 [1 to 6] | 1.5 [1 to 2] | 2 [1 to 4] | 2 [1 to 8]
  Day 15 (n=1,3,4,18): number analyzed (Participants) | 1 | 3 | 4 | 18
  Day 15 (n=1,3,4,18) | 1 [1 to 1] | 2 [1 to 4] | 1.04 [0.82 to 2] | 2 [0.98 to 6]
  Week 8 (n=2,0,0,2): number analyzed (Participants) | 2 | 0 | 0 | 2
  Week 8 (n=2,0,0,2) | 10.5 [10.3 to 10.7] |  |  | 4.75 [1.92 to 7.58]
  Week 12 (n=2,0,0,3): number analyzed (Participants) | 2 | 0 | 0 | 3
  Week 12 (n=2,0,0,3) | 18.8 [15.5 to 22.1] |  |  | 4.88 [0.92 to 23.3]
  Week 16 (n=1,1,0,1): number analyzed (Participants) | 1 | 1 | 0 | 1
  Week 16 (n=1,1,0,1) | 11.8 [11.8 to 11.8] | 23 [23 to 23] |  | 2.23 [2.23 to 2.23]
  Week 20 (n=1,0,1,1): number analyzed (Participants) | 1 | 0 | 1 | 1
  Week 20 (n=1,0,1,1) | 11.5 [11.5 to 11.5] |  | 0.42 [0.42 to 0.42] | 0.87 [0.87 to 0.87]

11. Secondary Outcome: AUC[0-8] of Dabrafenib and Derived Metabolites in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Area under the concentration-time curve from zero (pre-dose) 8 hours (AUC[0-8]) of Dabrafenib and derived metabolites were listed and summarized using descriptive statistics.
Time Frame: Day 1, Day 15, Week 8 (Dabrafenib derived metabolites), Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 8 | 19
h*ng/mL
  Dabrafenib @ D1 (n=3,4,8,19) | 8750 (70.1) | 8250 (134.8) | 6880 (54.3) | 5200 (77.2)
  Dabrafenib @ D15 (n=1,3,4,15): number analyzed (Participants) | 1 | 3 | 4 | 15
  Dabrafenib @ D15 (n=1,3,4,15) | 7300 (NA) — Only one participant analyzed | 7220 (93.5) | 3390 (223.0) | 5060 (57.5)
  Dabrafenib @ Wk12 (n=0,0,0,1): number analyzed (Participants) | 0 | 0 | 0 | 1
  Dabrafenib @ Wk12 (n=0,0,0,1) |  |  |  | 372 (NA) — Only one participant analyzed
  Dabrafenib @ Wk16 (n=0,1,0,0): number analyzed (Participants) | 0 | 1 | 0 | 0
  Dabrafenib @ Wk16 (n=0,1,0,0) |  | 593 (NA) — Only one participant analyzed |  |
  Dabrafenib @ Wk20 (n=0,1,0,0): number analyzed (Participants) | 0 | 1 | 0 | 0
  Dabrafenib @ Wk20 (n=0,1,0,0) |  | 1090 (NA) — Only one participant analyzed |  |
  GSK2167542 @ D1 (n=3,3,6,18): number analyzed (Participants) | 3 | 3 | 6 | 18
  GSK2167542 @ D1 (n=3,3,6,18) | 302 (26.9) | 75.4 (174.5) | 93.4 (70.5) | 52.6 (137.6)
  GSK2167542 @ D15 (n=1,3,4,14): number analyzed (Participants) | 1 | 3 | 4 | 14
  GSK2167542 @ D15 (n=1,3,4,14) | 1720 (NA) — Only one participant analyzed | 1960 (54.6) | 1900 (87.4) | 1490 (117.2)
  GSK2167542 @ Wk8 (n=1,2,0,1): number analyzed (Participants) | 1 | 2 | 0 | 1
  GSK2167542 @ Wk8 (n=1,2,0,1) | 506 (NA) — Only one participant analyzed | 624 (92.2) |  | 343 (NA) — Only one participant analyzed
  GSK2167542 @ Wk12 (n=1,2,0,1): number analyzed (Participants) | 1 | 2 | 0 | 1
  GSK2167542 @ Wk12 (n=1,2,0,1) | 260 (NA) — Only one participant analyzed | 250 (22.9) |  | 480 (NA) — Only one participant analyzed
  GSK2167542 @ Wk16 (n=2,2,0,1): number analyzed (Participants) | 2 | 2 | 0 | 1
  GSK2167542 @ Wk16 (n=2,2,0,1) | 331 (14.3) | 308 (128.2) |  | 538 (NA) — Only one participant analyzed
  GSK2167542 @ Wk20 (n=0,2,0,1): number analyzed (Participants) | 0 | 2 | 0 | 1
  GSK2167542 @ Wk20 (n=0,2,0,1) |  | 603 (163.3) |  | 460 (NA) — Only one participant analyzed
  GSK2285403 @ D1 (n=3,3,7,18): number analyzed (Participants) | 3 | 3 | 7 | 18
  GSK2285403 @ D1 (n=3,3,7,18) | 6610 (49.5) | 6730 (99.5) | 4440 (30.7) | 3090 (89.1)
  GSK2285403 @ D15 (n=1,3,4,14): number analyzed (Participants) | 1 | 3 | 4 | 14
  GSK2285403 @ D15 (n=1,3,4,14) | 4470 (NA) — Only one participant analyzed | 3510 (48.5) | 2130 (178.5) | 1970 (126.2)
  GSK2285403 @ Wk8 (n=1,2,0,1): number analyzed (Participants) | 1 | 2 | 0 | 1
  GSK2285403 @ Wk8 (n=1,2,0,1) | 61.6 (NA) — Only one participant analyzed | 443 (6273.4) |  | 156 (NA) — Only one participant analyzed
  GSK2285403 @ Wk12 (n=1,2,0,1): number analyzed (Participants) | 1 | 2 | 0 | 1
  GSK2285403 @ Wk12 (n=1,2,0,1) | 42.1 (NA) — Only one participant analyzed | 41.1 (1.9) |  | 255 (NA) — Only one participant analyzed
  GSK2285403 @ Wk16 (n=2,2,0,1): number analyzed (Participants) | 2 | 2 | 0 | 1
  GSK2285403 @ Wk16 (n=2,2,0,1) | 94.2 (170.6) | 96.6 (100.1) |  | 83.2 (NA) — Only one participant analyzed
  GSK2285403 @ Wk20 (n=0,2,0,1): number analyzed (Participants) | 0 | 2 | 0 | 1
  GSK2285403 @ Wk20 (n=0,2,0,1) |  | 104 (1.48) |  | 154 (NA) — Only one participant analyzed

12. Secondary Outcome: AUC[0-8] of Trametinib in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Area under the concentration-time curve from zero (pre-dose) 8 hours (AUC[0-8]) of Trametinib was listed and summarized using descriptive statistics.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 8 | 19
h*ng/mL
  Day 1 (n=3,3,8,19): number analyzed (Participants) | 3 | 3 | 8 | 19
  Day 1 (n=3,3,8,19) | 21.3 (12.6) | 22.3 (59.5) | 32.9 (42.2) | 16.4 (108.1)
  Day 15 (n=1,3,3,16): number analyzed (Participants) | 1 | 3 | 3 | 16
  Day 15 (n=1,3,3,16) | 141 (NA) — Only one participant analyzed | 134 (24.3) | 152 (24.9) | 111 (35.5)
  Week 8 (n=2,0,0,0): number analyzed (Participants) | 2 | 0 | 0 | 0
  Week 8 (n=2,0,0,0) | 73.6 (54.6) |  |  |
  Week 12 (n=2,0,0,1): number analyzed (Participants) | 2 | 0 | 0 | 1
  Week 12 (n=2,0,0,1) | 49.6 (67.1) |  |  | 74.6 (NA) — Only one participant analyzed
  Week 16 (n=1,1,0,0): number analyzed (Participants) | 1 | 1 | 0 | 0
  Week 16 (n=1,1,0,0) | 99.2 (NA) — Only one participant analyzed | 89.6 (NA) — Only one participant analyzed |  |
  Week 20 (n=1,0,0,0): number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 20 (n=1,0,0,0) | 90.4 (NA) — Only one participant analyzed |  |  |

13. Secondary Outcome: Ctau of Dabrafenib and Derived Metabolites in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Pre-dose (trough) concentration at the end of the dosing interval (Ctau) of Dabrafenib and derived metabolites were listed and summarized using descriptive statistics.
Time Frame: Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 27 | 38
ng/mL
  Dabrafenib @ D15 (n=2,4,27,38): number analyzed (Participants) | 2 | 4 | 27 | 38
  Dabrafenib @ D15 (n=2,4,27,38) | 36.7 (73.1) | 59.7 (691.6) | 65.8 (180.0) | 63.3 (138.6)
  Dabrafenib @ Wk8 (n=3,2,2,4): number analyzed (Participants) | 3 | 2 | 2 | 4
  Dabrafenib @ Wk8 (n=3,2,2,4) | 76.1 (132.8) | 343 (10622.8) | 65.8 (85.3) | 110 (1636.5)
  Dabrafenib @ Wk12 (n=3,4,1,4): number analyzed (Participants) | 3 | 4 | 1 | 4
  Dabrafenib @ Wk12 (n=3,4,1,4) | 169 (65.0) | 40.2 (132.1) | 361 (NA) — Only one participant analyzed | 381 (3566.2)
  Dabrafenib @ Wk16 (n=3,2,2,4): number analyzed (Participants) | 3 | 2 | 2 | 4
  Dabrafenib @ Wk16 (n=3,2,2,4) | 65.3 (190.1) | 36.7 (129.6) | 23.5 (621.7) | 187 (2138.5)
  Dabrafenib @ Wk20 (n=2,2,2,4): number analyzed (Participants) | 2 | 2 | 2 | 4
  Dabrafenib @ Wk20 (n=2,2,2,4) | 116 (203.6) | 38 (499.4) | 45.5 (2117.6) | 234 (4585.4)
  GSK2167542 @ D15 (n=2,4,27,38): number analyzed (Participants) | 2 | 4 | 27 | 38
  GSK2167542 @ D15 (n=2,4,27,38) | 202 (44.9) | 249 (26.4) | 237 (123.8) | 276 (90.3)
  GSK2167542 @ Wk8 (n=3,2,2,4): number analyzed (Participants) | 3 | 2 | 2 | 4
  GSK2167542 @ Wk8 (n=3,2,2,4) | 553 (72.9) | 312 (88.8) | 154 (5.5) | 129 (114.9)
  GSK2167542 @ Wk12 (n=3,4,1,4): number analyzed (Participants) | 3 | 4 | 1 | 4
  GSK2167542 @ Wk12 (n=3,4,1,4) | 171 (48.9) | 146 (21.0) | 134 (NA) — Only one participant analyzed | 378 (67.0)
  GSK2167542 @ Wk16 (n=3,2,2,4): number analyzed (Participants) | 3 | 2 | 2 | 4
  GSK2167542 @ Wk16 (n=3,2,2,4) | 138 (99.0) | 135 (79.4) | 100 (74.1) | 381 (63.1)
  GSK2167542 @ Wk20 (n=2,2,2,4): number analyzed (Participants) | 2 | 2 | 2 | 4
  GSK2167542 @ Wk20 (n=2,2,2,4) | 267 (21.3) | 269 (110.5) | 87.8 (9.5) | 254 (146.9)
  GSK2285403 @ D15 (n=2,4,27,38): number analyzed (Participants) | 2 | 4 | 27 | 38
  GSK2285403 @ D15 (n=2,4,27,38) | 62.7 (53.1) | 69.5 (226.7) | 52.3 (135.9) | 54.2 (136.8)
  GSK2285403 @ Wk8 (n=3,2,2,4): number analyzed (Participants) | 3 | 2 | 2 | 4
  GSK2285403 @ Wk8 (n=3,2,2,4) | 95.9 (119.1) | 221 (6687.0) | 76 (83.3) | 88 (1592.9)
  GSK2285403 @ Wk12 (n=3,4,1,4): number analyzed (Participants) | 3 | 4 | 1 | 4
  GSK2285403 @ Wk12 (n=3,4,1,4) | 93.3 (205.6) | 49.6 (126.3) | 275 (NA) — Only one participant analyzed | 264 (593.9)
  GSK2285403 @ Wk16 (n=3,2,2,4): number analyzed (Participants) | 3 | 2 | 2 | 4
  GSK2285403 @ Wk16 (n=3,2,2,4) | 76.6 (187.2) | 42.5 (59.0) | 32.7 (287.3) | 157 (666.6)
  GSK2285403 @ Wk20 (n=2,2,2,4): number analyzed (Participants) | 2 | 2 | 2 | 4
  GSK2285403 @ Wk20 (n=2,2,2,4) | 162 (156.0) | 46.4 (189.2) | 58.9 (1252.0) | 170 (411.9)

14. Secondary Outcome: Ctau of Trametinib in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Pre-dose (trough) concentration at the end of the dosing interval (Ctau) of Trametinib was listed and summarized using descriptive statistics.
Time Frame: Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 27 | 38
ng/mL
  Day 15 (n=2,4,27,38): number analyzed (Participants) | 2 | 4 | 27 | 38
  Day 15 (n=2,4,27,38) | 8.35 (23.4) | 11.8 (9.1) | 10.8 (36.9) | 9.98 (40.5)
  Week 8 (n=3,2,2,4): number analyzed (Participants) | 3 | 2 | 2 | 4
  Week 8 (n=3,2,2,4) | 7.37 (56.5) | 10.4 (NA) — Not estimable due to insufficient number of participants with events. | 9.58 (27.5) | 11.6 (224.2)
  Week 12 (n=3,4,1,4): number analyzed (Participants) | 3 | 4 | 1 | 4
  Week 12 (n=3,4,1,4) | 6.6 (46.7) | 8.39 (158.9) | 7.51 (NA) — Only one participant analyzed | 15.8 (78.7)
  Week 16 (n=3,2,2,4): number analyzed (Participants) | 3 | 2 | 2 | 4
  Week 16 (n=3,2,2,4) | 4.55 (114.3) | 8.92 (33.1) | 6.66 (8.1) | 19.4 (68.1)
  Week 20 (n=2,2,2,4): number analyzed (Participants) | 2 | 2 | 2 | 4
  Week 20 (n=2,2,2,4) | 6.91 (78.8) | 8.67 (16.4) | 6.81 (1.6) | 7.28 (317.3)

15. Secondary Outcome: Ctau of Panitumumab in the Triple Combination (D+T+P)
Description: Serial blood samples were collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples were collected every 4 weeks up to and including Week 20 on study. Pre-dose (trough) concentration at the end of the dosing interval (Ctau) of Panitumumab was listed and summarized using descriptive statistics.
Time Frame: Day 15, Week 4, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 24 | 34
ng/mL
  Day 15 (n=3,3,24,34): number analyzed (Participants) | 3 | 3 | 24 | 34
  Day 15 (n=3,3,24,34) | 11100 (52.8) | 25600 (53.2) | 9860 (99.0) | 21300 (64.5)
  Week 4 (n=0,0,20,26): number analyzed (Participants) | 0 | 0 | 20 | 26
  Week 4 (n=0,0,20,26) |  |  | 18100 (73.4) | 37000 (52.9)
  Week 8 (n=3,2,1,4): number analyzed (Participants) | 3 | 2 | 1 | 4
  Week 8 (n=3,2,1,4) | 46300 (37.7) | 29900 (66.7) | 19300 (NA) — Only one participant analyzed | 27900 (57.7)
  Week 12 (n=3,4,0,3): number analyzed (Participants) | 3 | 4 | 0 | 3
  Week 12 (n=3,4,0,3) | 34700 (53.1) | 36100 (51.6) |  | 31700 (85.8)
  Week 16 (n=3,2,1,3): number analyzed (Participants) | 3 | 2 | 1 | 3
  Week 16 (n=3,2,1,3) | 14000 (326.7) | 56400 (4.8) | 29400 (NA) — Only one participant analyzed | 25200 (85.5)
  Week 20 (n=2,2,2,3): number analyzed (Participants) | 2 | 2 | 2 | 3
  Week 20 (n=2,2,2,3) | 24400 (NA) — Not estimable due to insufficient number of participants with events. | 35400 (4.2) | 23800 (NA) — Not estimable due to insufficient number of participants with events | 40700 (46.3)

16. Secondary Outcome: Apparent Base Clearance (CL0/F) and Apparent Maximum Inducible Clearance at Steady State (CLIND,SS/F) of Dabrafenib in the Triple Combination (D+T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The apparent base clearance (CL0/F) and apparent maximum inducible clearance at steady state (CLIND,SS/F) of Dabrafenib estimated with the PopPK model are summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: All subjects who received at least one dose of dabrafenib in Part 1, 2A and 2B and provided an evaluable PK profile. All trametinib and dabrafenib concentration-time data were combined and included in a population PK analysis that examined the influence of demographics on the PK of study treatment.
Measure: Number (95% Confidence Interval); unit: L/h
Groups:
- Part 1+2A+2B - Triple Combination (D+T+P): All Participants With PK Data: Participants in Part 1+2A+2B - Triple combination (D+T+P) of the study (all doses) with available pharmacokinetic data
Arm/Group | Part 1+2A+2B - Triple Combination (D+T+P): All Participants With PK Data
Number analyzed (Participants) | 90
L/h
  Apparent base clearance (CL0/F) | 16.7 [15.3 to 18.1]
  Apparent maximum inducible clearance at steady state (CLIND,SS/F) | 18.6 [17.7 to 19.5]

17. Secondary Outcome: Effect of Combination With Trametinib on Apparent Maximum Inducible Clearance at Steady State of Dabrafenib in the Triple Combination (D+T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The effect of combination with trametinib on apparent maximum inducible clearance at steady state (CLIND,SS/F) (CLCOMBO) of Dabrafenib estimated with the PopPK model is summarized in this record.
  The parameter in question is a covariate that describes the effect of Effect of combination with trametinib on apparent maximum inducible clearance: the number denoting the effect means that the including trametinib will decrease the apparent maximum inducible clearance as opposed to when dabrafenib is administered alone.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: no unit of measure
Arm/Group | Part 1+2A+2B - Triple Combination (D+T+P): All Participants With PK Data
Number analyzed (Participants) | 90
no unit of measure | 0.625 [0.578 to 0.672]

18. Secondary Outcome: Oral Volume of Distribution (V/F) of Dabrafenib in the Triple Combination (D+T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The oral volume of distribution (V/F) of Dabrafenib of Dabrafenib estimated with the PopPK model is summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Liter (L)
Arm/Group | Part 1+2A+2B - Triple Combination (D+T+P): All Participants With PK Data
Number analyzed (Participants) | 90
Liter (L) | 58.5 [53.6 to 63.4]

19. Secondary Outcome: Absorption Rate Constant (Ka) of Dabrafenib in the Triple Combination (D+T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The absorption rate constant (Ka) of Dabrafenib estimated with the PopPK model is summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: 1/h
Arm/Group | Part 1+2A+2B - Triple Combination (D+T+P): All Participants With PK Data
Number analyzed (Participants) | 90
1/h | 1.22 [1.06 to 1.38]

20. Secondary Outcome: Cmax of Trametinib in the Double Combination (T+P)
Description: as for outcome 8
Time Frame: Day 1, Day 15, Week 12, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W
Number analyzed (Participants) | 1 | 2 | 0
ng/mL
  Day 1 (n=0,2,0): number analyzed (Participants) | 0 | 2 | 0
  Day 1 (n=0,2,0) |  | 1.53 (164.4) |
  Day 15 (n=1,2,0) | 22.9 (NA) — Only one participant analyzed | 12 (47.1) |
  Week 12 (n=1,0,0): number analyzed (Participants) | 1 | 0 | 0
  Week 12 (n=1,0,0) | 19.3 (NA) — Only one participant analyzed |  |
  Week 20 (n=1,0,0): number analyzed (Participants) | 1 | 0 | 0
  Week 20 (n=1,0,0) | 29.9 (NA) — Only one participant analyzed |  |

21. Secondary Outcome: Tmax of Trametinib in the Double Combination (T+P)
Description: as for outcome 10
Time Frame: Day 1, Day 15, Week 12, Week 20
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W
Number analyzed (Participants) | 1 | 2 | 0
Hour (hr)
  Day 1 (n=0,2,0): number analyzed (Participants) | 0 | 2 | 0
  Day 1 (n=0,2,0) |  | 2.5 [1 to 4] |
  Day 15 (n=1,2,0) | 4 [4 to 4] | 3 [2 to 4] |
  Week 12 (n=1,0,0): number analyzed (Participants) | 1 | 0 | 0
  Week 12 (n=1,0,0) | 4.07 [4.07 to 4.07] |  |
  Week 20 (n=1,0,0): number analyzed (Participants) | 1 | 0 | 0
  Week 20 (n=1,0,0) | 5.72 [5.72 to 5.72] |  |

22. Secondary Outcome: AUC[0-t] of Trametinib in the Double Combination (T+P)
Description: Serial blood samples will be collected pre-dose and post-dose on Day 1, Day 15 and pre-dose on Day 21 in the first 28 days of dosing. In the continuation period, blood samples will be collected every 4 weeks up to and including Week 20 on study. Area under the concentration-time curve from zero (pre-dose) the time of the last quantifiable concentration (AUC[0-t]) of Trametinib was listed and summarized using descriptive statistics.
Time Frame: Day 1, Day 15, Week 12, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W
Number analyzed (Participants) | 1 | 2 | 0
h*ng/mL
  Day 1 (n=0,2,0): number analyzed (Participants) | 0 | 2 | 0
  Day 1 (n=0,2,0) |  | 2.78 (718.3) |
  Day 15 (n=1,2,0) | 81 (NA) — Only one participant analyzed | 38.4 (56.5) |
  Week 12 (n=1,0,0): number analyzed (Participants) | 1 | 0 | 0
  Week 12 (n=1,0,0) | 78.6 (NA) — Only one participant analyzed |  |
  Week 20 (n=1,0,0): number analyzed (Participants) | 1 | 0 | 0
  Week 20 (n=1,0,0) | 171 (NA) — Only one participant analyzed |  |

23. Secondary Outcome: Ctau of Trametinib in the Double Combination (T+P)
Description: as for outcome 14
Time Frame: Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W
Number analyzed (Participants) | 9 | 15 | 14
ng/mL
  Day 15 (n=9,15,14) | 11 (19.8) | 9.44 (34.0) | 11.2 (38.8)
  Week 8 (n=4,6,7): number analyzed (Participants) | 4 | 6 | 7
  Week 8 (n=4,6,7) | 4.71 (251.5) | 3.36 (154.1) | 7.66 (116.3)
  Week 12 (n=4,5,6): number analyzed (Participants) | 4 | 5 | 6
  Week 12 (n=4,5,6) | 4.54 (368.1) | 7.28 (62.7) | 4.26 (98.4)
  Week 16 (n=1,2,1): number analyzed (Participants) | 1 | 2 | 1
  Week 16 (n=1,2,1) | 8.37 (NA) — Only one participant analyzed | 5.07 (16.1) | 1.49 (NA) — Only one participant analyzed
  Week 20 (n=2,1,1): number analyzed (Participants) | 2 | 1 | 1
  Week 20 (n=2,1,1) | 13.1 (170.4) | 5.48 (NA) — Only one participant analyzed | 10.7 (NA) — Only one participant analyzed

24. Secondary Outcome: Ctau of Panitumumab in the Double Combination (T+P)
Description: as for outcome 15
Time Frame: Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W
Number analyzed (Participants) | 9 | 11 | 11
ng/mL
  Day 15 (n=9,11,11) | 16000 (47.4) | 17400 (44.0) | 8160 (65.9)
  Week 8 (n=4,5,6): number analyzed (Participants) | 4 | 5 | 6
  Week 8 (n=4,5,6) | 25300 (18.9) | 10000 (233.2) | 9570 (40.8)
  Week 12 (n=5,2,4): number analyzed (Participants) | 5 | 2 | 4
  Week 12 (n=5,2,4) | 13600 (80.7) | 31700 (NA) — Not estimable due to insufficient number of participants with events. | 5210 (24.7)
  Week 16 (n=3,0,0): number analyzed (Participants) | 3 | 0 | 0
  Week 16 (n=3,0,0) | 3510 (3526.0) |  |
  Week 20 (n=2,1,0): number analyzed (Participants) | 2 | 1 | 0
  Week 20 (n=2,1,0) | 11800 (NA) — Not estimable due to insufficient number of participants with events. | NA (NA) — Only one participant analyzed |

25. Secondary Outcome: Apparent Base Clearance (CL0/F) and Apparent Maximum Inducible Clearance at Steady State (CLIND,SS/F) of Dabrafenib in the Double Combination (T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The apparent base clearance (CL0/F) and apparent maximum inducible clearance at steady state (CLIND,SS/F) dabrafenib estimated with the PopPK model are summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: All subjects who received at least one dose of dabrafenib in Part 4A and 4B and provided an evaluable PK profile. All trametinib and dabrafenib concentration-time data were combined and included in a population PK analysis that examined the influence of demographics on the PK of study treatment.
Measure: Number (95% Confidence Interval); unit: L/h
Groups:
- Part 4A+4B - Double Combination (T+P): All Participants With PK Data: Participants in Part 4A+4B of the study (all doses) with available pharmacokinetic data
Arm/Group | Part 4A+4B - Double Combination (T+P): All Participants With PK Data
Number analyzed (Participants) | 49
L/h
  Apparent base clearance (CL0/F) | 16.7 [15.3 to 18.1]
  Apparent maximum inducible clearance at steady state (CLIND,SS/F) | 18.6 [17.7 to 19.5]

26. Secondary Outcome: Oral Volume of Distribution (V/F) of Dabrafenib in the Double Combination (T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Dabrafenib can be described using a two-compartment model with a delayed 1st order absorption (Alag1, Ka) and an inducible elimination (CL/F) that consists of a base clearance (constant over time, CL0/F) and a dose- and time-dependent inducible clearance (CLind/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of dabrafenib. The oral volume of distribution (V/F) of Dabrafenib estimated with the PopPK model is summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Liter (L)
Arm/Group | Part 4A+4B - Double Combination (T+P): All Participants With PK Data
Number analyzed (Participants) | 49
Liter (L) | 58.5 [53.6 to 63.4]

27. Secondary Outcome: Absorption Rate Constant (Ka) of Dabrafenib in the Double Combination (T+P) Estimated With a PopPK Model
Description: as for outcome 19
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: 1/h
Arm/Group | Part 4A+4B - Double Combination (T+P): All Participants With PK Data
Number analyzed (Participants) | 49
1/h | 1.22 [1.06 to 1.38]

28. Secondary Outcome: Apparent Clearance (CL/F) of Trametinib in the Double Combination (T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Trametinib can be described using a two-compartment model with dual sequential 1st order absorption (Ka1, Ka2) and 1st order elimination (CL/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of trametinib. The apparent clearance (CL/F) of Trametinib estimated with the PopPK model is summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: L/h
Arm/Group | Part 4A+4B - Double Combination (T+P): All Participants With PK Data
Number analyzed (Participants) | 49
L/h | 5.07 [4.82 to 5.32]

29. Secondary Outcome: Apparent Central Volume (V/F) of Trametinib in the Double Combination (T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Trametinib can be described using a two-compartment model with dual sequential 1st order absorption (Ka1, Ka2) and 1st order elimination (CL/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of trametinib. The apparent central volume (V/F) of Trametinib estimated with the PopPK model is summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: Liter (L)
Arm/Group | Part 4A+4B - Double Combination (T+P): All Participants With PK Data
Number analyzed (Participants) | 49
Liter (L) | 184 [158 to 210]

30. Secondary Outcome: Absorption Rate Constant 1 (Ka1) and Absorption Rate Constant 2 (Ka2) of Trametinib in the Double Combination (T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Trametinib can be described using a two-compartment model with dual sequential 1st order absorption (Ka1, Ka2) and 1st order elimination (CL/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of trametinib. The absorption rate constant 1 (Ka1) and absorption rate constant 2 (Ka2) of Trametinib estimated with the PopPK model are summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: 1/h
Arm/Group | Part 4A+4B - Double Combination (T+P): All Participants With PK Data
Number analyzed (Participants) | 49
1/h
  Absorption rate constant 1 (Ka1) | 0.134 [0.075 to 0.193]
  Absorption rate constant 2 (Ka2) | 1.55 [1.05 to 2.05]

31. Secondary Outcome: Time When Ka1 Transitions to Ka2 of Trametinib in the Double Combination (T+P) Estimated With a PopPK Model
Description: The population pharmacokinetic (PopPK) model of Trametinib can be described using a two-compartment model with dual sequential 1st order absorption (Ka1, Ka2) and 1st order elimination (CL/F). The PopPK analysis examined the influence of demographics (i.e., weight) on the pharmacokinetics of trametinib. The time when Ka1 transitions to Ka2 of Trametinib estimated with the PopPK model is summarized in this record.
Time Frame: Day 1, Day 15, Week 8, Week 12, Week 16, Week 20
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: hour (h)
Arm/Group | Part 4A+4B - Double Combination (T+P): All Participants With PK Data
Number analyzed (Participants) | 49
hour (h) | 0.404 [0.344 to 0.464]

32. Secondary Outcome: Change in Levels of Proteins/Ribonucleic Acid (RNA)
Description: H-score or "Histo-score" measures cell membrane immunohistochemistry staining intensity in a fixed field. Membrane staining is categorized as 1+, 2+, or 3+. Minimum score is 0, maximum score is 300 (no subscale values are reported). H-score values themselves are not considered to be better or worse - measurements for levels of proteins/ribonucleic acid (RNA) are surrogate for MAPK pathway activity. Low values = low pathway activity. High values = high pathway activity. Changes in mean phosphorylated-ERK (pERK) and phosphorylated ribosomal protein S6 (pS6) H-score from baseline indicate changes in MAPK pathway activity that may be associated with treatment arms. A positive change from baseline suggests increased pathway activity. A negative change from baseline suggests decreased pathway activity. Total score is calculated as follows: [1 x (% cells 1+) + 2 x (% cells 2+) + 3 x (% cells 3+)].
Time Frame: Baseline, Day 15
Population: All treated population. Parameter information at baseline of patients with two different baseline were excluded. Day 15 included post-baseline information between study day 13 - 18.
Measure: Mean (Standard Deviation); unit: H-Score
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 36 | 50 | 11 | 10 | 10 | 2 | 10 | 10 | 20
H-Score
  pERK H score: Baseline (BL) (n=1,3,13,15,4,4,5,1,4,4,11): number analyzed (Participants) | 1 | 3 | 13 | 15 | 4 | 4 | 5 | 1 | 4 | 4 | 11
  pERK H score: Baseline (BL) (n=1,3,13,15,4,4,5,1,4,4,11) | 60.0 (NA) — Only 1 participant analyzed | 195.7 (14.01) | 140.7 (96.51) | 148.7 (83.46) | 114.3 (60.31) | 255.3 (33.72) | 209.2 (89.95) | 145.0 (NA) — Only 1 participant analyzed | 146.3 (71.81) | 188.8 (33.26) | 163.9 (80.84)
  pERK H score: D15 (n=1,2,10,14,4,4,6,1,4,4,11): number analyzed (Participants) | 1 | 2 | 10 | 14 | 4 | 4 | 6 | 1 | 4 | 4 | 11
  pERK H score: D15 (n=1,2,10,14,4,4,6,1,4,4,11) | 210.0 (NA) — Only 1 participant analyzed | 30.5 (27.58) | 73.8 (59.93) | 82.6 (78.16) | 40.0 (39.16) | 52.5 (65.89) | 131.3 (36.04) | 100.0 (NA) — Only 1 participant analyzed | 155.0 (54.47) | 171.0 (76.18) | 149.2 (81.68)
  pERK H score @ change from BL @ D15 (n=1,2,10,13,4,4,5,1,4,4,10): number analyzed (Participants) | 1 | 2 | 10 | 13 | 4 | 4 | 5 | 1 | 4 | 4 | 10
  pERK H score @ change from BL @ D15 (n=1,2,10,13,4,4,5,1,4,4,10) | 150.0 (NA) — Only 1 participant analyzed | -158.0 (18.38) | -62.9 (71.41) | -66.0 (56.12) | -74.3 (44.92) | -202.8 (74.41) | -77.2 (97.77) | -45.0 (NA) — Only 1 participant analyzed | 8.8 (110.78) | -17.8 (102.67) | -14.7 (77.91)
  pS6 H score: Baseline (BL) (n=1,3,13,15,4,4,6,1,4,4,10): number analyzed (Participants) | 1 | 3 | 13 | 15 | 4 | 4 | 6 | 1 | 4 | 4 | 10
  pS6 H score: Baseline (BL) (n=1,3,13,15,4,4,6,1,4,4,10) | 175.0 (NA) — Only 1 participant analyzed | 209.3 (77.50) | 143.7 (80.48) | 102.3 (75.55) | 194.0 (132.70) | 193.8 (83.40) | 180.8 (75.59) | 40.0 (NA) — Only 1 participant analyzed | 51.0 (51.48) | 65.5 (50.71) | 202.8 (86.14)
  pS6 H score: D15 (n=1,2,10,14,4,4,6,1,4,4,11): number analyzed (Participants) | 1 | 2 | 10 | 14 | 4 | 4 | 6 | 1 | 4 | 4 | 11
  pS6 H score: D15 (n=1,2,10,14,4,4,6,1,4,4,11) | 260.0 (NA) — Only 1 participant analyzed | 60.0 (70.71) | 59.7 (78.21) | 68.0 (76.64) | 67.8 (76.81) | 98.5 (110.15) | 64.3 (73.21) | 40.0 (NA) — Only 1 participant analyzed | 44.8 (53.92) | 72.8 (88.31) | 130.1 (75.70)
  pS6 H score @ change from BL @ D15 (n=1,2,10,13,4,4,6,1,4,4,9): number analyzed (Participants) | 1 | 2 | 10 | 13 | 4 | 4 | 6 | 1 | 4 | 4 | 9
  pS6 H score @ change from BL @ D15 (n=1,2,10,13,4,4,6,1,4,4,9) | 85.0 (NA) — Only 1 participant analyzed | -107.5 (31.82) | -68.1 (61.49) | -27.2 (66.65) | -126.3 (101.27) | -95.3 (88.35) | -116.5 (103.16) | -50.0 (NA) — Only 1 participant analyzed | -6.3 (15.28) | 7.3 (101.26) | -70.4 (67.19)

33. Secondary Outcome: Part 3: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) using RECIST 1.1
Time Frame: as for outcome 2
Population: as for outcome 3
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Part 3: Duration of Response (DoR)
Description: as for outcome 4
Time Frame: as for outcome 2
Population: as for outcome 3
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Part 3: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time to death due to any cause.
Time Frame: From study treatment start date until date of of death from any cause, assessed up to approximately 90 months
Population: as for outcome 3
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) mBRAF: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P) Anti-EGFR: TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

36. Secondary Outcome: Part 3: Number of Participants With Treatment Emergent Adverse Events
Description: The distribution of adverse events (AE) will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From study treatment start date till 30 days safety follow-up, assessed up to approximately 90 months
Population: as for outcome 3
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

37. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 2454 days (treatment duration ranged from 1 to 2424 days).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approximately 7 years. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: up to 2454 days (on-treatment), up to approximately 7 years (study duration)
Population: Clinical database population; all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
Number analyzed (Participants) | 3 | 4 | 36 | 50 | 13 | 20 | 20 | 20
Participants
  On-treatment deaths | 0 | 0 | 3 | 2 | 1 | 2 | 0 | 0
  Post-treatment deaths | 3 | 4 | 25 | 42 | 11 | 15 | 17 | 16
  All deaths | 3 | 4 | 28 | 44 | 12 | 17 | 17 | 16

ADVERSE EVENTS:
Time Frame: On-treatment Adverse events (AEs) and serious AEs (including the All-Cause Mortality data table) are presented from first dose of study treatment until last dose of study treatment plus 30 days post treatment, for a maximum duration of 2454 days (treatment duration ranged from 1 to 2424 days).
Description: Any sign or symptom that occurs during the study treatment and 30 days post treatment follow up.
  Maximum exposure to study treatments = 2424 days in the Trametinib (T) plus Dabrafenib (D) plus Panitumumab (P) Triplet Combination (T+D+P), 508 days in the Trametinib (T) plus Panitumumab (P) Doublet Combination (T+P) and 652 days in the Dabrafenib (D) plus Panitumumab (P) Doublet Combination (D+P).
Arm/Group | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 3/36 | 2/50 | 1/13 | 2/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 21/36 | 28/50 | 6/13 | 10/20 | 9/20 | 6/20
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 36/36 | 50/50 | 13/13 | 20/20 | 20/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W (N=3) | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W (N=4) | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W (N=36) | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W (N=50) | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W (N=13) | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W (N=20) | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W (N=20) | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5 | 1 | 0 | 2 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 3 | 8 | 1 | 2 | 1 | 4
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Splenic abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinoma (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 4.8MG/KG Q2W (N=3) | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 1.5MG QD, PAN 6MG/KG Q2W (N=4) | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 4.8MG/KG Q2W (N=36) | Part 1+2A+2B - Triple Combination (T+D+P): DAB 150MG BID, TRA 2MG QD, PAN 6MG/KG Q2W (N=50) | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 6MG/KG Q2W (N=13) | Part 4A+4B - Double Combination (T+P): TRA 1.5MG QD, PAN 6MG/KG Q2W (N=20) | Part 4A+4B - Double Combination (T+P): TRA 2MG QD, PAN 4.8MG/KG Q2W (N=20) | Part 1+2A - Double Combination (D+P): DAB 150MG BID, PAN 6MG/KG Q2W (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 8 | 18 | 2 | 7 | 5 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 4 | 2 | 2 | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Trichomegaly (Eye disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 3 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 4 | 6 | 5 | 4 | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 6 | 4 | 0 | 0 | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 11 | 8 | 2 | 3 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 21 | 31 | 10 | 15 | 13 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 4 | 5 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 5 | 2 | 0 | 0 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 22 | 27 | 7 | 7 | 6 | 9
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 8 | 9 | 0 | 7 | 6 | 2
Vomiting (Gastrointestinal disorders) | 3 | 3 | 16 | 18 | 7 | 7 | 3 | 6
Asthenia (General disorders) | 1 | 2 | 6 | 5 | 3 | 5 | 6 | 3
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 6 | 3 | 1 | 2 | 1 | 5
Fatigue (General disorders) | 1 | 1 | 18 | 25 | 7 | 2 | 4 | 9
Influenza like illness (General disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 3 | 3 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 6 | 8 | 2 | 4 | 3 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 0 | 10 | 12 | 3 | 1 | 5 | 1
Peripheral swelling (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 16 | 26 | 4 | 7 | 9 | 4
Xerosis (General disorders) | 1 | 0 | 2 | 3 | 2 | 2 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 2 | 4 | 5 | 1 | 3 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 14 | 12 | 0 | 4 | 4 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pustule (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 3 | 3 | 1 | 3 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 4 | 5 | 2 | 4 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 5 | 8 | 2 | 5 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 6 | 2 | 2 | 2 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 2 | 5 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 2 | 2 | 0 | 3 | 2
Globulins increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 7 | 11 | 3 | 1 | 1 | 4
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 13 | 22 | 4 | 7 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2 | 5 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 6 | 8 | 3 | 0 | 4 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 3 | 2 | 2 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 12 | 3 | 4 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 8 | 18 | 6 | 7 | 3 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 5 | 2 | 2 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 2 | 1 | 0 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 4 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 3 | 2 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 1 | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4 | 1 | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 5 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 7 | 9 | 2 | 2 | 1 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 6 | 1 | 3 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 4 | 2 | 1 | 0 | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 4 | 2 | 1 | 3 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 3 | 1 | 0 | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 7 | 4 | 1 | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5 | 1 | 1 | 1 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 3 | 25 | 27 | 7 | 7 | 10 | 12
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 20 | 27 | 5 | 8 | 6 | 7
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 0 | 1 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 9 | 5 | 1 | 1 | 3 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 2 | 2 | 1 | 1 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4 | 1 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 5 | 1 | 1 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 14 | 8 | 2 | 4 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 8 | 20 | 5 | 8 | 6 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 8 | 4 | 3 | 0 | 3 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 1 | 9 | 10 | 2 | 3 | 5 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 2 | 2 | 1 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 3 | 6 | 0 | 2 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT01750918/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT01750918/SAP_001.pdf